CLINICAL TRIAL: NCT06520514
Title: Safety, Tolerability, and Relative Bioavailability of a Single Dose of Spesolimab Via Two Subcutaneous Modes of Delivery in Healthy Subjects (Mono-centric, Randomised, Parallel Group Design)
Brief Title: A Study to Test How Well Healthy People Tolerate Spesolimab When Given in 2 Different Ways
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1368-0151; 2023-510448-20-00 (Registry Identifier: CTIS); U1111-1301-8808 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reference group (Active Comparator): Reference treatment using the standard administration mode
  Interventions: Drug: Spesolimab
- Test 1 group (Experimental): Treatment 1 using the test administration mode
  Interventions: Drug: Spesolimab
- Test 2 group (Experimental): Treatment 2 using the test administration mode
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Spesolimab
  Other Names: BI 655130

SUMMARY:
The main objectives of this trial is to investigate the safety and tolerability of a single dose of spesolimab administered in 2 different ways in healthy subjects.

ELIGIBILITY:
Inclusion Criteria :

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests.
* Age of 18 to 50 years (inclusive).
* Body mass index (BMI) of 18.5 to 30.0 kg/m^2 (inclusive).
* Signed and dated written informed consent in accordance with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Women of childbearing potential (WOCBP) must meet any of the following criteria for a highly effective contraception starting from at least 30 days before the administration of trial medication until 16 weeks after the injection/infusion of trial medication:

  * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal),
  * Use of progestogen-only hormonal contraception that inhibits ovulation (oral, injectable or implantable),
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS),
  * Bilateral tubal occlusion/ ligation,
  * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm in ejaculate) and provided that partner is the sole sexual partner of the woman of childbearing potential trial participant,
  * Complete abstinence (refraining from heterosexual intercourse) is considered a highly effective method of contraception only if it is in line with the preferred and usual lifestyle of the trial participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to trial investigational medicinal product, and withdrawal (coitus interruptus) are not acceptable.

Exclusion Criteria :

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator.
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders.
* History of relevant orthostatic hypotension, fainting spells, or blackouts.
* Participants with relevant chronic infections as determined by the investigator, including active or latent tuberculosis, Human Immunodeficiency Virus (HIV) or viral hepatitis. The corresponding laboratory tests will be performed during screening. In case of a positive hepatitis C antibody test, a positive reflex testing for Hepatitis C RNA (Ribonucleic Acid) PCR (polymerase chain reaction) is considered positive. For hepatitis B, exclusion criterion is met with either a positive Hepatitis B surface antigen or a positive Hepatitis B virus (HBV) DNA (Deoxyribonucleic Acid) PCR (HBV DNA PCR is done in case of positive Hepatitis core antibody and negative Hepatitis B surface antigen.).

Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event | Up to day 120

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | Up to day 120
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to day 120
Cmax (maximum measured concentration of the analyte in plasma) | Up to day 120

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com